CLINICAL TRIAL: NCT01609595
Title: An Open Label Academic Phase 2 Study of SDMB in Subjects in Thailand With Beta Thalassemia Intermedia
Brief Title: Study of SDMB (2,2 Dimethylbutyrate, Sodium Salt) in Beta Thalassemia Intermedia in Thailand
Acronym: ST20-P2T
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Mahidol University (Other)
Responsible Party: Principal Investigator, Susan P. Perrine, Sponsor Investigator, Boston University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST20-P2T; HQK-1001-Thal P2 (Other: HemaQuest)
Record Dates: First submitted 2012-04-25; First posted 2012-06-01 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Beta Thalassemia Intermedia
Keywords: Thalassemia; Anemia; Fetal hemoglobin
MeSH Terms: conditions — beta-Thalassemia; Thalassemia; Anemia | interventions — 2,2-dimethylbutyric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Study drug treatment
  Interventions: Drug: sodium 2,2 dimethylbutyrate

INTERVENTIONS:
Drug: sodium 2,2 dimethylbutyrate — Oral capsule, dose 20 mg/kg/day, daily, for 26 weeks
  Other Names: HQK-1001, ST20

SUMMARY:
Beta thalassemia intermedia is an inherited blood disease caused by molecular mutations which reduce the beta globin protein chain of adult hemoglobin A, the protein in red blood cells which carries oxygen throughout the body. Beta thalassemias cause progressively severe anemia, widespread organ damage, and often require blood transfusions. There is no FDA approved therapeutic to treat the underlying cause of beta thalassemia. Fetal hemoglobin is another type of endogenous hemoglobin which can replace the reduced beta globin protein, reduce the anemia, and even abolish transfusion requirements. This type of hemoglobin is normally suppressed in infancy.

Sodium 2,2 dimethylbutyrate (ST20, or HQK-1001) is a small molecule which stimulates production of fetal hemoglobin in nonhuman primates and in human patients in Phase I/II trials.

This is a Phase 2 open-label trial to evaluate the ability of this oral therapeutic to reduce anemia in patients with beta thalassemia intermedia, when administered once daily for 26 weeks. All participants will receive the study drug.

DETAILED DESCRIPTION:
This trial will:

1. Determine the proportion of patients in which treatment with the study drug results in an increase in total hemoglobin by 1.5 g/dl above baseline levels when administered for 26 weeks in Thai patients with beta thalassemia intermedia, including Hemoglobin E beta thalassemia.
2. Determine the number and proportion of participants in whom treatment with the study drug results in an increase in fetal hemoglobin.
3. Determine the number of participants who have adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Beta Thalassemia Intermedia
* Splenectomized
* Average of two Hgb levels between 6.0 and 9.0 g/dl

Exclusion Criteria:

* Red blood cell transfusion within 3 months of study drug initiation
* Enlarged spleen
* Use of hydroxyurea within 6 months
* QT Segment corrected (QTc)> 450 msec (men) or 470 msec (women) on screening ECG
* Use of iron chelating agents within 7 days of first dose
* Alanine Transaminase(ALT)> 4 times the upper limit of normal
* Use of erythropoiesis stimulating agents (ESAs) within 90 days of first dose
* serum creatinine > 1.5 mg/dL

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-03; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The number of participants in which an increase in total hemoglobin of at least 1.5 g/dl above average baseline occurs with study drug treatment. | Within 30 weeks, including 26 weeks of dosing with the study drug
  Baseline hemoglobin levels will be determined by averaging 2 values prior to administration of the study drug.
  The number of participants in which an increase in total hemoglobin of at least 1.5 g/dL above baseline occurs will be determined.

SECONDARY OUTCOMES:
The proportion of participants in which an increase in fetal hemoglobin occurs above the subjects' averaged baseline levels. | Within 30 weeks, including 26 weeks of study drug administration
  Tests of fetal hemoglobin will be obtained at two times prior to administration of the study drug and will be averaged. Laboratory tests of fetal hemoglobin will be assessed monthly during the study drug administration for 26 weeks, as a biomarker of drug activity.

CONTACTS AND LOCATIONS:
Overall Officials: Suthat Fuchareon, MD, Principal Investigator — Thalassemia Research Centre, Mahidol University
Locations (1):
- Mahidol University Thalassemia Research Centre, Nakhonpathom, Thailand

REFERENCES:
- [Background] Perrine SP, Castaneda SA, Chui DH, Faller DV, Berenson RJ, Siritanaratku N, Fucharoen S. Fetal globin gene inducers: novel agents and new potential. Ann N Y Acad Sci. 2010 Aug;1202:158-64. doi: 10.1111/j.1749-6632.2010.05593.x. PMID 20712788
- [Background] Perrine SP, Wargin WA, Boosalis MS, Wallis WJ, Case S, Keefer JR, Faller DV, Welch WC, Berenson RJ. Evaluation of safety and pharmacokinetics of sodium 2,2 dimethylbutyrate, a novel short chain fatty acid derivative, in a phase 1, double-blind, placebo-controlled, single-dose, and repeat-dose studies in healthy volunteers. J Clin Pharmacol. 2011 Aug;51(8):1186-94. doi: 10.1177/0091270010379810. Epub 2011 Mar 21. PMID 21422239